CLINICAL TRIAL: NCT00957034
Title: A Placebo-controlled Study to Determine the Efficacy and Safety of 300 and 450 µg/Day Transdermal Testosterone in Female Patients With Low Ejection Fraction and Symptomatic Heart Failure
Brief Title: Assessing the Safety/Efficacy of Transdermal Testosterone in Female Patients With Symptomatic Heart Failure
Acronym: CORDELIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to difficult patient enrollment.
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009015
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2011-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo (Placebo Comparator): placebo patch
  Interventions: Drug: placebo
- 300 µg/day testosterone (Experimental): 300 micrograms/day transdermal testosterone patch
  Interventions: Drug: testosterone
- 450 µg/day testosterone (Experimental): 450 micrograms/day transdermal testosterone patch
  Interventions: Drug: testosterone

INTERVENTIONS:
Drug: placebo — placebo patch
  Arms: placebo
Drug: testosterone — 300 or 450 micrograms/day transdermal testosterone patch
  Arms: 300 µg/day testosterone; 450 µg/day testosterone

SUMMARY:
Heart failure (HF) is a complex condition resulting from structural or functional heart diseases that impair the ability of the heart to fill with or pump out blood. The main manifestations of HF are shortness of breath and tiredness which may limit the ability to exercise or perform simple daily physical activities such as walking. Heart disease leading to HF is associated with reduced muscle mass and reduced strength and low blood levels of testosterone; a hormone normally produced by the human (male and female) body. Recent studies have shown improvements of symptoms and ability to exercise in patients with heart failure receiving testosterone.

This is a placebo controlled study to determine the efficacy and safety of low dose testosterone (300 and 450 microgram/day) delivered by a transdermal system (patch) in women with significant HF.

ELIGIBILITY:
Inclusion Criteria:

* Female 50 years of age or older; post-menopausal (≥ 12 Mo/ from last menstruation)
* Documented left ventricular ejection fraction (LVEF) of 20-40% within 90 days prior to the baseline visit
* History of HF for more than 90 days and a diagnosis of symptomatic HF (Class III NYHA) for at least 30 days prior to the baseline visit
* Ambulatory (i.e., able to walk without assistance of another person or device such as cane or walker)

Exclusion Criteria:

* Neuromuscular or rheumatologic conditions that limit the to their ability to improve walking distance
* Pulmonary edema or multiorgan failure or cardiogenic shock within 30 days prior to the baseline visit
* Congenital heart disease, infiltrative myocardial disease
* Unstable angina or myocardial infarction within 30 days prior to the baseline visit
* Undiagnosed abnormal genital bleeding
* History of breast cancer, breast surgery, or breast disease contraindicating estrogen/hormone therapy
* Polycystic ovary syndrome or any other condition known to be adversely affected by testosterone treatment
* Resting heart rate > 120 bpm
* Systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg
* Known or suspected hypersensitivity or allergy to any adhesive or to any of the components of the testosterone transdermal system (TTS)
* Use of SERMS, SARMS, SPRMs, tibolone, testosterone, estrogen, progesterone agonists and antagonists or taking any prescription and over the counter medications/ nutraceuticals (eg, phyto-estrogens) that may have anabolic or steroid hormonal effects within 30 days prior to the baseline visit
* Use of marketed or investigational oral, sub-lingual, topical, transdermal injectable, or vaginal androgen therapy including dehydroepiandrosterone (DHEA) at any time within 3 months prior to the baseline visit
* Use of systemic corticosteroids within 30 days prior to the baseline visit (acute use for fewer than 7 days is acceptable)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Brum, MD, Study Director — Procter and Gamble
Locations (16):
- United States (16):
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Lakewood, California
  - Research Site, Riverside, California
  - Research Site, Stamford, Connecticut
  - Research Site, Melbourne, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Savannah, Georgia
  - Research Site, Munster, Indiana
  - Research Site, Brooklyn, New York
  - Research Site, Wilmington, North Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Germantown, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 month trial, screening started 22 Sep 2009 and ended 24 Mar 2010.
Period: Overall Study
Arm/Group | Placebo | 300 µg/Day Testosterone | 450 µg/Day Testosterone
Started | 6 | 4 | 7
Completed | 0 | 0 | 1
Not Completed | 6 | 4 | 6
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Sponsor Terminated Study | 6 | 1 | 5
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 300 µg/Day Testosterone | 450 µg/Day Testosterone | Total
Number analyzed (Participants) | 6 | 4 | 7 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 70.3 (6.2) | 69.8 (5.0) | 74.3 (9.0) | 71.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 7 | 17
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Six Minute Walking Test (6MWT), Meters
Description: Measurement of distance walked as fast as possible on a hard flat pathway in six minutes
Time Frame: Baseline and Day 180
Population: No statistical analysis performed due to early termination of the study. Study was stopped prior to any subjects reaching a timepoint for efficacy assessment. Safety results were available and recorded in the interim.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | 300 µg/Day Testosterone | 450 µg/Day Testosterone
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Percent Change From Baseline in Severity of Heart Failure (HF) as Measured by New York Heart Association (NYHA) Classification
Description: Class I: Cardiac disease w/o limitation of physical activity. Class II: Cardiac disease resulting in slight limitation of physical activity. Comfortable at rest; ordinary activity results in fatigue, palpitation, dyspnea or anginal pain. Class III: Cardiac disease resulting in marked limitation of physical activity. Comfortable at rest; less than ordinary activity causes fatigue, palpitation, dyspnea or anginal pain. Class IV: Cardiac disease resulting in inability to carry on any physical activity w/o discomfort. Symptoms present at rest. Any physical activity increases discomfort.
Time Frame: Baseline and Day 180
Population: as for outcome 1
Measure: Number; unit: Percent Change
Arm/Group | Placebo | 300 µg/Day Testosterone | 450 µg/Day Testosterone
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Mortality or Hospitalizations
Description: Composite endpoint - patients who were hospitalized or died during the trial.
Time Frame: Baseline and Day 180
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | 300 µg/Day Testosterone | 450 µg/Day Testosterone
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Percent Change Minnesota Living With Heart Failure Questionnaire (MLHFQ) Overall Score and Domain Scores
Description: Minnesota Living with Heart Failure Questionnaire assessing how much heart failure affects life during previous month. Three scales measuring physical dimension (8 items, score 0-40), emotional dimension (5 items, score 0-25) and overall score (all 21 items, score 0-105). Eight separate items measure social & economic impairments included as part of overall score.
Time Frame: Baseline and Day 180
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | 300 µg/Day Testosterone | 450 µg/Day Testosterone
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Percent Change Patient Global Assessment of Heart Failure Status
Description: Four global questions classifying improvement or deterioration in heart failure - Since your last clinic vist, has there been any change in activity limitation / symptoms / emotions / overall quality of life, related to your heart failure? Scale -7/very great deal worse, -6 great deal worse, -5 good deal worse, -4 moderately worse, -3 somewhat worse, -2 a little worse, -1 hardly any worse/almost the same, 0 no change, 1 hardly better/almost the same, 2 little better, 3 somewhat better, 4 moderately better, 5 good deal better, 6 great deal better, 7 very great deal better.
Time Frame: Baseline and Day 180
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | 300 µg/Day Testosterone | 450 µg/Day Testosterone
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Percent Change Physician Global Assessment of Heart Failure Status
Description: Physician rates improvement or deterioration in heart failure: Scale -7/very great deal worse, -6 great deal worse, -5 good deal worse, -4 moderately worse, -3 somewhat worse, -2 a little worse, -1 hardly any worse/almost the same, 0 no change, 1 hardly better/almost the same, 2 little better, 3 somewhat better, 4 moderately better, 5 good deal better, 6 great deal better, 7 very great deal better.
Time Frame: Baseline and Day 180
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | 300 µg/Day Testosterone | 450 µg/Day Testosterone
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Six-month treatment period.
Arm/Group | Placebo | 300 µg/Day Testosterone | 450 µg/Day Testosterone
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/4 | 2/7
Other Adverse Events (participants affected / at risk) | 4/6 | 2/4 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | 300 µg/Day Testosterone (N=4) | 450 µg/Day Testosterone (N=7)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | 300 µg/Day Testosterone (N=4) | 450 µg/Day Testosterone (N=7)
Application Site Reaction (General disorders) | 1 (1) | 1 (1) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tendon Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Breast Mass (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less